CLINICAL TRIAL: NCT00966706
Title: PEXG (Cisplatin, Epirubicin, Capecitabine, Gemcitabine) Versus PDXG (Cisplatin, Docetaxel, Capecitabine, Gemcitabine) in Locally Advanced or Metastatic Pancreatic Adenocarcinoma: A Randomized Phase II Trial
Brief Title: Cisplatin, Capecitabine, Gemcitabine and Epirubicin or Docetaxel for Patients With Stage III or IV Pancreatic Cancer
Acronym: PACT-9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000642240; SRSI-PACT-9 (Other: IRCCS San Raffaele); 2005-002586-36 (EudraCT Number)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Cisplatin; Docetaxel; Epirubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive cisplatin, gemcitabine hydrochloride, and docetaxel on days 1 and 15, and capecitabine on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride
- Arm II (Experimental): Patients receive cisplatin, gemcitabine hydrochloride, and epirubicin hydrochloride on days 1and 15, and capecitabine on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine — Given systemically
  Other Names: XELODA
Drug: cisplatin — Given systemically
  Other Names: Cisplatino-TEVA
Drug: docetaxel — Given systemically
  Other Names: TAXOTERE
  Arms: Arm I
Drug: epirubicin hydrochloride — Given systemically
  Other Names: FARMARUBICINA
  Arms: Arm II
Drug: gemcitabine hydrochloride — Given systemically
  Other Names: GEMZAR

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, capecitabine, gemcitabine hydrochloride, epirubicin hydrochloride, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether cisplatin, capecitabine, and gemcitabine hydrochloride are more effective when given together with epirubicin hydrochloride or docetaxel in treating patients with advanced or metastatic pancreatic cancer.

PURPOSE: This randomized phase II trial is studying the side effects of giving cisplatin, capecitabine, and gemcitabine hydrochloride together with epirubicin hydrochloride compared with giving cisplatin, capecitabine, and gemcitabine hydrochloride together with docetaxel and to see how well it works in treating patients with stage III or stage IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess 6-months progression-free survival of patients with stage III or IV adenocarcinoma of the pancreas treated with cisplatin, capecitabine, gemcitabine hydrochloride (PXG) and epirubicin hydrochloride vs PXG and docetaxel.
* Evaluate the activity and toxicity of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I (PEXG): Patients receive cisplatin, gemcitabine hydrochloride, and docetaxel on days 1 and 15, and capecitabine on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (PGDX): Patients receive cisplatin, gemcitabine hydrochloride, and epirubicin hydrochloride on days 1and 15, and capecitabine on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients may then undergo surgery if the tumor becomes resectable.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic adenocarcinoma of the pancreas

  * Stage III or IV disease
* Measurable disease
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Adequate bone marrow, liver, and kidney function
* Not pregnant or nursing
* No other malignancies within the past 5 years except surgically treated carcinoma in situ of the cervix, and basal or squamous cell carcinoma of the skin
* No multiple severe diseases that can compromise study safety, including any of the following:

  * Cardiac failure
  * Myocardial infarction within the past 4 months
  * Cardiac arrhythmia
  * History of psychiatric disabilities

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for pancreatic cancer
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6-months | every 2 months during therapy; every 3 months thereafter
  CT scan

SECONDARY OUTCOMES:
Overall survival | monthly
Response rate | every 2 months during therapy; every 3 months thereafter
  CT scan
Toxicity | every 2 weeks during therapy
  outpatient visit

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy